CLINICAL TRIAL: NCT06019338
Title: A Study to Validate a Diary Developed by Noema Pharma That Will be Used for Future Trigeminal Neuralgia Clinical Research Studies to Capture Pain Dimensions.
Brief Title: A Study to Validate a Pain Diary for Patient With Trigeminal Neuralgia
Status: Completed | Type: Observational
Sponsor: Noema Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: NOE-PRO-001
Record Dates: First submitted 2022-05-01; First posted 2023-08-31 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2023-11

CONDITIONS: Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pain Diary use — Validation of a pain diary specifically designed to capture pain dimensions of Trigeminal Neuralgia

SUMMARY:
The aim of the study is to establish the validity of a patient reported diary in TN . The following objectives have been identified:

1. To generate evidence to support diary content validity by performing qualitative research studies with TN patients and Healthcare Professionals (HCPs).
2. To provide further support to the diary, sensitivity to change, known groups validity (ability to differentiate between severity groups), and construct validity.

DETAILED DESCRIPTION:
This study will engage up to 20 participants with TN through patient associations or HCPs. The study will be conducted in English Speaking countries.

The study comprises the following parts :

* Participants Recruitment
* Completion of the Diary
* Qualitative interviews with participants
* Analysis of qualitative research to assess content validity
* Secondary analysis as a workshop with a panel of experts to finalize the diary The diary will be provided to each participant and to HCPs. Participants will be requested to follow the instructions, use the diary and provide their feedback on the diary.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female aged of 40 years or more.
* Must be able to read, write, and speak English to complete the consent process and participate in an interview.
* Able and willing to provide consent for participation in the study, and to allow the study team to access their data entries including audio or video recordings. - - Participant with a current or previous diagnosis of TN
* Willing to participate in up to 30 minutes remote interviews or in-person interview (this interview will be recorded by the HCP)
* Committ to fill in the diary according to the HCP instruction

Exclusion Criteria:

* Not applicable

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients or former patients with diagnosed trigeminal neuralgia
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-11-20 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Measure of pain associated with Trigeminal Neuralgia | 2 weeks
  Use of the TN Pain questionnaire to measure the pain associated with trigeminal neuralgia
Concept elicitation of the diary content | 1 day
  During an interview, assess if the questionnaire is comprehensive, clear and correctly captures patients experience

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director, Study Director — Noema Pharma AG
Locations (2):
- Kainzen Centre, La Jolla, California, United States
- ULC Research, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No